CLINICAL TRIAL: NCT05650853
Title: Study of the Biomechanical Anatomy of Ejaculation
Brief Title: Exploration of eJaculatory Anatomy Concept Study (EJAC Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Dr Vincent Misrai, Principal Investigator, MD, Clinique Pasteur
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-A01594-39
Record Dates: First submitted 2022-11-10; First posted 2022-12-14 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Ejaculatory Dysfunction
MeSH Terms: conditions — Ejaculatory Dysfunction | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study intervention (Experimental): Transrectal ultrasound and Urethroscopy
  Interventions: Other: Transrectal ultrasound; Other: Urethroscopy

INTERVENTIONS:
Other: Transrectal ultrasound — Examinations for observation of the pre, per and post-ejaculatory phases
Other: Urethroscopy — Examinations for observation of the pre, per and post-ejaculatory phases

SUMMARY:
Ejaculatory dysfunctions (ED) are an important cause of postoperative dissatisfaction, which lead to a decrease in the intensity of orgasms in 50% of patients. ED is a cause for concern for almost a third of patients who need surgery. Surgical techniques have been developed to limit the occurrence of postoperative ED, but their results remain heterogeneous.

There are very few studies on the biomechanical anatomy of ejaculation. Ejaculation is a complex phenomenon involving different structures and in particular the Veru Montanum. This is the key element in the emission of ejaculate within the prostatic urethra. In addition, there is a structure located in the resection zone of the prostate adenoma. It has therefore been suggested that its resection was a primary source of ED.

A single observational study carried out in by Gil Vernet et al in 1994 evaluated on a single healthy 18-year-old volunteer the ejaculatory mechanism of expulsion using an endorectal probe recording the movements of the prostate, the bladder neck and of the proximal urethra during ejaculation.

A contemporary study of the biomechanics of the ejaculatory expulsion phase could confirm and improve understanding of the involvement of anatomical structures. The results of our study aim to adapt surgical techniques aimed at limiting the risk of postoperative ED.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated subject or beneficiary of a social security scheme
* Subject agreeing to participate and having signed the free, informed consent.

Exclusion Criteria:

* Subject with ejaculatory dysfunction
* Subject with urinary dysfunction
* History of urinary or penile surgery
* Subject with untreated urinary tract infection
* History of chronic prostatitis
* Pathology making it impossible to introduce the endorectal probe or the ureteroscope
* History of colorectal inflammatory disease
* Recent intake (within 30 days) of drugs known to interfere with ejaculation
* History of intolerance or allergy to any of the drugs used in the study
* Subject participating in another clinical study
* Adults under guardianship, curatorship or other legal protection; deprived of liberty by judicial or administrative decision; Hospitalized without consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Peri-urethral muscle contraction | At Day 0
  Qualitative description of peri-urethral muscle contraction according to ultrasound videos analysis
Urethra, bladder neck and prostate movements | At Day 0
  Qualitative description of movements of the urethra, bladder neck and prostate according to ultrasound videos analysis
Sperm flow within the prostatic urethra | At Day 0
  Qualitative description of sperm flow within the prostatic urethra according to ultrasound videos analysis
Spermatic fluid via the ejaculatory ducts | At Day 6
  Qualitative description of the expulsion and flow of spermatic fluid via the ejaculatory ducts according to urethroscopy videos analysis
Veru montanum mobility and urethral contraction. | At Day 6
  Qualitative description of veru montanum mobility and urethral contraction according to urethroscopy videos analysis

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pradère, MD, Study Director — Clinique La Croix du Sud; Eric Bruguière, MD, Study Director — Clinique Pasteur; Vincent Misraï, MD, Study Director — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: No